CLINICAL TRIAL: NCT05599022
Title: Randomized Assessment of the Efficacy of Transcutaneous Magnetic Stimulation in Patients With Ventricular Tachycardia Storm
Brief Title: Randomized Assessment of TcMS for VT Storm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 852176
Record Dates: First submitted 2022-10-24; First posted 2022-10-31 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Sham Stimulation (Placebo Comparator): With the coil directed away from the patient, 600 pulses of TcMS will be delivered at minimal energy output.
  Interventions: Device: Magnetic Stimulation
- Low Frequency TcMS (Active Comparator): With the coil directed at the stellate ganglion, 60 minutes of 1Hz stimulation will be delivered targeting the stellate ganglion.
  Interventions: Device: Magnetic Stimulation
- Theta Burst Stimulation TcMS (Active Comparator): With the coil directed at the stellate ganglion, 600 pulses of continuous theta burst stimulation will be delivered targeting the stellate ganglion.
  Interventions: Device: Magnetic Stimulation

INTERVENTIONS:
Device: Magnetic Stimulation — Transcutaneous Magnetic Stimulation

SUMMARY:
Three-arm randomized clinical trial comparing two strategies of TcMS to sham stimulation in patients with VT storm. The hypothesis of the study is that TcMS will reduce the burden of VT in the 24 hours after randomization compared to sham stimulation and that TcMS with theta burst stimulation (TBS) will be more effective at reducing VT burden than low frequency TcMS.

ELIGIBILITY:
Inclusion Criteria:

* ≥3 episodes of sustained VT or appropriate ICD therapies within 24 hours despite the use of at least one antiarrhythmic drug

Exclusion Criteria:

* Plan for catheter ablation of VT in the next 24 hours
* Pregnancy
* Contraindication to TcMS (i.e. implantable ventricular assist device, metal implanted in the head or neck [except the mouth], implanted medication pumps, cochlear implant, implanted brain stimulator, ocular implant, history of malignancy in the neck)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
VT Burden (24 hours) | 24 hours after randomization
  Number of episodes of sustained ventricular tachycardia

SECONDARY OUTCOMES:
VT burden (72 hours) | 72 hours after randomization
  Number of episodes of sustained ventricular tachycardia
Freedom from VT | 24 hours after randomization
  Freedom from sustained VT
Blood Pressure | Immediately before and after stimulation
  Change in mean arterial blood pressure
Heart Rate | Immediately before and after stimulation
  Change in heart rate
Pain | Immediately after stimulation
  Pain at site of stimulation (0-10 scale)
Lead sensing | Immediately before and after stimulation
  Change in implantable device lead sensing
Lead threshold | Immediately before and after stimulation
  Change in implantable device lead pacing threshold
Lead impedance | Immediately before and after stimulation
  Change in implantable device lead pacing impedance

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No